CLINICAL TRIAL: NCT04914988
Title: Pain Management in Geriatric Hip Fracture Patients With Ultrasound-guided Continuous Fascia Iliaca Compartment Block
Brief Title: Continuous Fascia Iliaca Compartment Block in Geriatric Hip Fracture
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suwimon Tangwiwat, Department of Anesthesiology, Mahidol University
Other Study IDs: Si 113/2018
Record Dates: First submitted 2021-05-26; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Hip Fractures; Acute Pain Due to Trauma
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The patient with hip fracture who has Numerical Rating Scale (NRS) ≥ 5 at rest or on movement will be indicated for USG FICB at Emergency Department or patient's ward.

The aim of this prospective observation study was evaluated the efficacy and complications of cFICB in adult hip fracture preoperatively.

DETAILED DESCRIPTION:
The Enhance Recovery Program of pain management in geriatric hip fracture has been set up as a part of fast track at Siriraj Hospital since September 2017. The ultrasound-guided (USG) fascia iliaca compartment block (FICB) is routinely offered to patients with a hip fracture by acute pain service (APS) anesthesiologist. The patient with hip fracture who has Numerical Rating Scale (NRS) ≥ 5 at rest or on movement will be indicated for USG FICB.

The aim of this prospective observation study was evaluated the efficacy and complications of cFICB in adult hip fracture preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patient age equal or more than 65 years old
* patient with acute hip fracture within 7 days
* patient with NRS ≥ 5

Exclusion Criteria:

* patient refusal
* history of local anesthetic allergy
* inability to communicate or cognitive dysfunction
* multiple fracture involvement

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Acute hip fracture in elderly
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
numerical rating scale at rest | Change from baseline numerical rating scale at 30 minutes post-block
  numerical rating scale 0-10 (0=no pain, 10=worst pain)
numerical rating scale during movement | Change from baseline numerical rating scale at 30 minutes post-block
  numerical rating scale 0-10 (0=no pain, 10=worst pain)

SECONDARY OUTCOMES:
Numerical rating scale during movement | Within 48 hours postoperative
  numerical rating scale 0-10 (0=no pain, 10=worst pain)
Rate of complications of continuous fascia iliaca compartment analgesia | Within 48 hours postoperative
  local anesthetic systemic toxicity, leakage, infection
Duration of hospital admission | from hospital admission until hospital discharge, an average of 1 week
  number of days
Number of participants with morbidity and mortality | 6 weeks after hospital discharge
  myocardial disease, deep vein thrombosis, delirium, death

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] White SM, Moppett IK, Griffiths R, Johansen A, Wakeman R, Boulton C, Plant F, Williams A, Pappenheim K, Majeed A, Currie CT, Grocott MP. Secondary analysis of outcomes after 11,085 hip fracture operations from the prospective UK Anaesthesia Sprint Audit of Practice (ASAP-2). Anaesthesia. 2016 May;71(5):506-14. doi: 10.1111/anae.13415. Epub 2016 Mar 4. PMID 26940645
- [Result] Guay J, Parker MJ, Gajendragadkar PR, Kopp S. Anaesthesia for hip fracture surgery in adults. Cochrane Database Syst Rev. 2016 Feb 22;2(2):CD000521. doi: 10.1002/14651858.CD000521.pub3. PMID 26899415
- [Result] Orosz GM, Magaziner J, Hannan EL, Morrison RS, Koval K, Gilbert M, McLaughlin M, Halm EA, Wang JJ, Litke A, Silberzweig SB, Siu AL. Association of timing of surgery for hip fracture and patient outcomes. JAMA. 2004 Apr 14;291(14):1738-43. doi: 10.1001/jama.291.14.1738. PMID 15082701
- [Result] Birnbaum K, Prescher A, Hessler S, Heller KD. The sensory innervation of the hip joint--an anatomical study. Surg Radiol Anat. 1997;19(6):371-5. doi: 10.1007/BF01628504. PMID 9479711
- [Result] Guay J, Parker MJ, Griffiths R, Kopp S. Peripheral nerve blocks for hip fractures. Cochrane Database Syst Rev. 2017 May 11;5(5):CD001159. doi: 10.1002/14651858.CD001159.pub2. PMID 28494088
- [Result] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544
- [Result] Ftouh S, Morga A, Swift C; Guideline Development Group. Management of hip fracture in adults: summary of NICE guidance. BMJ. 2011 Jun 21;342:d3304. doi: 10.1136/bmj.d3304. No abstract available. PMID 21693526